CLINICAL TRIAL: NCT05208164
Title: My ESSENCE - Mindfulness to Reduce Stress, Improve SIeep, and Reduce Cardiovascular Risk in African-Americans With Type 2 Diabetes
Brief Title: My ESSENCE - A Research Study on Mindfulness for African-Americans With Type 2 Diabetes
Acronym: E-RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Alana Biggers, Primary Investigator, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2019-1433; 1K01HL149775 (NIH)
Record Dates: First submitted 2021-12-10; First posted 2022-01-26 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Type 2 Diabetes; Sleep; Stress
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Group A will be assigned as the intervention group and Group B will be assigned as the usual care group. During the pilot RCT, Group A will run in parallel with Group B.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Meditation Classes (Experimental): 8 mindfulness classes: Participants will engage in 8 two-hour mind and body practice classes over 8 weeks in-person or online (during the pandemic). You will receive compensation for your participation and a yoga mat. You will need to wear comfortable clothing. These sessions can be done sitting in chair, sitting on the floor, or standing.
  Text messaging., in between classes you will receive text messages to encourage mind and body practices at home. Text messaging may appear as the following:
  1.Do you have time to meditate right now? Yes or No. 2.Did you practice your mindfulness today? Yes or no. 3.Remember to wind down this evening and do not drink any caffeinated beverages 4 hours before bed.
  Interventions: Behavioral: Mindfunlness Meditation
- Usual Care (No Intervention)

INTERVENTIONS:
Behavioral: Mindfunlness Meditation — Sleep monitoring, mental health promotion and active enrollment/engagement in self-described coping mechanisms
  Arms: Mindfulness Meditation Classes

SUMMARY:
The proposed research and training will allow Dr. Alana Biggers to obtain critical research skills and study a mindfulness meditation program designed to improve sleep and reduce stress in African-American adults with diabetes. If effective, this program may reduce the risk of cardiovascular disease among African-Americans with type 2 diabetes who are at high risk of cardiovascular disease.

DETAILED DESCRIPTION:
African-Americans have disproportionate rates of cardiovascular disease (CVD) in the US. African-Americans with type 2 diabetes (T2DM) have twice the risk than non-Hispanic whites for developing CVD. Poorer sleep and greater chronic psychological stress may contribute to this additional risk. Consequently, African-Americans have worse glycemic control among those with diabetes and higher CVD risk. One promising approach to improving CVD risk in African-Americans is mindfulness meditation (MM). MM can potentially reduce cardiovascular risk through attention control, emotional regulation, and self-awareness. The overall purpose of this K01 training grant is for Dr. Alana Biggers to obtain research training and develop skills needed to become an independent investigator, and use those skills to adapt and evaluate an established MM curriculum. The specific aims are to: (1) adapt and refine an established MM curriculum for African-Americans with T2DM and incorporate text messaging; (2) conduct an 8-week, pilot randomized, controlled trial of the adapted curriculum with up to 100 African-Americans with T2DM(goal of 68 for study completion); and (3) explore the impact of the intervention on cardiometabolic risk factors (blood pressure, glycosylated hemoglobin, and lipid profile) and inflammatory biomarkers (C-reactive protein, interleukin-6, and tumor necrosis factor α). Primary outcomes will include sleep quality and perceived stress evaluated at baseline, 8, and 16 weeks. The proposed research design consists of a pilot study, utilizes mixed-methods research, and involves both primary data collection and analysis. Participants will be randomized 1:1 to either the MM intervention or control. Patients will be assigned to fill cohorts so that those in intervention group will attend MM classes together. A cohort represents a group of 10-12 subjects enrolled within a 1-month time period. MM classes will guide participants in learning and implementing MM practices over 8 weeks. Data collection will occur at baseline, 8 weeks (completion of MM sessions), and 16 weeks. The 16-week data assessment will evaluate MM practice beyond the MM class structure to assess for sustainability.

This K01 training grant will provide Dr. Biggers career-building activities to further develop skills and a knowledge base in quantitative and qualitative methodology, health disparities research, and mobile health (mHealth)/behavioral health strategies in minority populations. With the guidance of an interdisciplinary mentorship team and institutional support, Dr. Biggers will receive the necessary assistance and training to work toward her long-term career goal of being an independent researcher with expertise in health disparities, mixed-methods, and mHealth behavioral research.

ELIGIBILITY:
Inclusion Criteria

* Self-identifies as African American or Black
* Diagnosis of type 2 diabetes
* Valid address in greater Chicagoland area
* Mobile phone with unlimited text-messaging
* Mobile device (smartphone, tablet, or computer) with the ability to connect to the internet if remote online delivery
* Availability to participate in mindfulness class either in-person or online
* Age 21-75

Exclusion Criteria

* Untreated obstructive sleep apnea (OSA)
* Severe insomnia, narcolepsy, or REM sleep related disorder
* Major cognitive impairments or psychiatric disorder
* Alcohol or drug abuse
* Limited English proficiency
* Inability to send/receive text messages
* Currently engaging in mindfulness practice

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Sleep Quality | Change from baseline at 8 and 16 weeks.
  Will use Pittsburgh Sleep Quality Index (PSQI). PSQI has a minimum score of 0 (better) and maximum of 21 (worse). Score > 5 is considered poor quality sleep.
Perceived Stress | Change from baseline at 8 and 16 weeks.
  Will use Perceived Stress Scale. Scale has a minimum value of 0, and maximum value of 40. Scores from 0-13 are considered low stress, 14-26 are moderate, and 27-40 are high perceived stress.
Sleep Disturbances | Change from baseline at 8 and 16 weeks
  Will use Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance Short Form 8b. Scores are reported as T-scores, with 28.9 being the minimum value, and 76.5 being the maximum. Higher scores indicate greater sleep disturbances.
Sleep Impairment | Change from baseline at 8 and 16 weeks
  Will use Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Related Impairment Short Form 8a.Scores are reported as T-scores, with 30.0 being the minimum value, and 80.1 being the maximum. Higher scores indicate greater sleep impairment.

SECONDARY OUTCOMES:
Cardiovascular Risk | Change from baseline at 8 weeks
  Fasting lipid profile (total cholesterol, HDL, LDL and triglycerides) and blood pressure will be combined to estimate 10 year cardiovascular risk using the American College of Cardiology Atherosclerotic Cardiovascular Disease (ACC ASCVD) Risk Estimator Plus Calculator.
Hemoglobin A1c | Change from baseline at 8 weeks.
  Will use HbgA1c as a measure for determining cardiovascular risk.
Inflammatory Markers | Change from baseline at 8 and 16 weeks
  IL-6, CRP, TNF-alpha

CONTACTS AND LOCATIONS:
Overall Officials: Alana Biggers, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No